CLINICAL TRIAL: NCT05324085
Title: Aerobic Exercise for Cognitive Functioning in Patients With Substance Use Disorder: a Randomized Controlled Trial
Brief Title: Aerobic Exercise for Cognitive Functioning in Patients With Substance Use Disorder
Acronym: SO_CogEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Lade Behandlingssenter, Blå Kors (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 171845; 3253020430 (Other Grant/Funding Number: Central Norway Regional Health Authority)
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Substance Abuse; Cognitive Dysfunction
Keywords: Exercise therapy; High-intensity interval training
MeSH Terms: conditions — Substance-Related Disorders; Cognitive Dysfunction | interventions — High-Intensity Interval Training; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention group (Experimental): Participants will undergo supervised treadmill exercise three times each week for eight weeks, in addition to treatment as usual (TAU).
  Interventions: Behavioral: High-intensity interval training; Behavioral: Treatment as usual
- Control group (Other): Participants will undergo TAU. The content of TAU is broadly individualized but most often includes various forms of group therapy, psychotherapy, psychoeducation and physical activity. The physical activity schedule for the patients typically includes gym-based exercises, individualized by preference of each patient, and various outdoors activities, four times per week all together.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: High-intensity interval training — Supervised exercise intervention, three times a week for eight weeks.
  Other Names: HIIT
  Arms: Exercise intervention group
Behavioral: Treatment as usual — The content of TAU is broadly individualized but most often includes various forms of group therapy, psychotherapy, psychoeducation and physical activity. The physical activity schedule for the patients typically includes gym-based exercises, individualized by preference of each patient, and various outdoors activities, four times per week all together.

SUMMARY:
Impaired cognitive function is common among patients with substance use disorder (SUD). This is particularly related to executive functions (EF), which includes abilities like decision-making, consequence analysis and impulse/self-control. EF is recognized as an important determinant of treatment outcome as it is associated with dropout rate, attendance to therapy sessions and absence of relapse following treatment termination. Exercise seem to improve cognitive/executive functions, particularly in individuals with cognitive impairments. Aerobic exercise also affects signaling substances and growth factors known to inhibit neural degeneration, and improves cerebral insulin sensitivity and blood flow, contributing to improved brain function. There is a lack of knowledge regarding how to improve EF in SUD patients, and whether such improvements can benefit other parts of the treatment, such as psychotherapy. Aerobic exercise is a well-recognized and cost-effective intervention for cardiovascular and metabolic health, with promising effects on cognitive/executive functions. A randomized controlled trial will be carried out to investigate the effects of aerobic exercise on EF, molecular markers of neuroplasticity and brain function, and treatment outcome in SUD patients. The investigators expect to achieve new knowledge regarding cognitive impairment among SUD patients and to what extent aerobic exercise can improve cognitive abilities and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed substance use disorder (SUD) by ICD-10
* Being in residential inpatient treatment for SUD at Lade Addiction Treatment Center

Exclusion Criteria:

* Recent participation in regular aerobic high-intensity interval training (HIIT)
* Admissions shorter than 12 weeks
* Pregnant
* History of brain injury (except concussions)
* Any acute or chronic somatic or psychiatric condition (e.g. heart disease or psychosis) or a medication that would limit the ability to participate in the exercise training and testing procedures, or any of the other assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change in executive function (EF) | 8 weeks
  Change in executive function assessed with Behavior Rating Inventory of ExecutiveFunction, Adult (BRIEF-A). BRIEF-A is a 75-item standardized questionnaire appraising EFs in real-life situations. It incorporates self-reported cognitive characteristics and collects subjective information about the ability to maintain appropriate control of emotional responses and behavior.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) score | 8 weeks
  MoCA is a brief neuropsychological assessment to evaluate cognitive function in various domains (i.e. visuospatial/executive abilities, naming, memory, attention, language, abstraction, and orientation). This assessment takes about 10 minutes to perform. Maximum score is 30, but scores from 26 and above is considered normal.
Change in Stroop test score | 8 weeks
  Stroop is a widely used and validated test evaluate attention and impulse control. This particular test allow 90 seconds to solve as many problems as possible. Each correct answer provides one point, while incorrect answers are subtracted from the total score.
Change in Digit Span test performance | 8 weeks
  The Digit Span test is an assessment of working memory, using rows of numbers that should be memorized. Each correct answer provides one point with the following sequence being one digit longer than the previous. The test has no limit on time or upper score, but only allows three mistakes before ending.
Altered serum concentration of Brain Derived Neurotrophic Factor (BDNF) | 8 weeks
  BDNF is a biochemical marker of neurocognitive/neuroprotective mechanisms that can be measured in human serum
Altered serum concentration of Klotho | 8 weeks
  Klotho is a biochemical marker of neurocognitive/neuroprotective mechanisms that can be measured in human serum
Altered serum concentration of glycosylphosphatidylinositol-specific phospholipase D1 (Gpld1) | 8 weeks
  Gpld1 is a biochemical marker of neurocognitive/neuroprotective mechanisms that can be measured in human serum
Altered serum concentration of interleukin 6 (IL6) | 8 weeks
  IL6 is a muscle-secreted protein known to affect neurocognitive/neuroprotective mechanisms
Change in maximal cardiorespiratory fitness | 8 weeks
  Maximal cardiorespiratory fitness will be measured as oxygen uptake by cardiopulmonary exercise testing on a treadmill, by inclined walking or running on a treadmill
Change in mental distress | 8 weeks
  Alterations in mental distress will be assessed using the validated brief questionnaire Symptom Checklist-10 (SCL-10)
Change in substance use | 8 weeks
  Change in substance use will be assessed using a simple self-report questionnaire
Change in substance craving | 8 weeks
  Change in substance use will be assessed using a simple Visual Analogue Scale ranging from 0 (no craving) to 10 (severe craving)
Change in quality of life | 8 weeks
  Quality of life will be assessed with a brief version of the World Health Organization Quality of Life assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mats P Mosti, PhD, Principal Investigator — Department of Research and Development, St. Olavs University Hospital
Locations (1):
- Lade Behandlingssenter, Blåkors, Trondheim, Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Plan in progress

REFERENCES:
- [Derived] Haberstroh C, Weider S, Flemmen G, Loe H, Andersson HW, Hallgren M, Mosti MP. The effect of high-intensity interval training on cognitive function in patients with substance use disorder: Study protocol for a two-armed randomized controlled trial. Front Sports Act Living. 2022 Dec 9;4:954561. doi: 10.3389/fspor.2022.954561. eCollection 2022. PMID 36570498